CLINICAL TRIAL: NCT07020169
Title: Artificial Intelligence-Driven 3D Kidney Model for Real-Time Augmented Reality and Surgical Navigation in Minimally Invasive (Robotic/Laparoscopic) Partial Nephrectomy: A Prospective Validation Study
Brief Title: Using 3D Kidney Model Based on Artificial Intelligence to Assist Partial Nephrectomy: A Prospective Validation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shao Pengfei (Other)
Collaborators: Southeast University, China (Other)
Responsible Party: Sponsor-Investigator, Shao Pengfei, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-309
Record Dates: First submitted 2025-05-24; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Cancer
Keywords: partial nephrectomy; Articicial Intelligence; Intraoperative Real-Time Navigation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Surgical Approaches (No Intervention): perform conventional laparoscopic or robotic-assisted surgical approaches
- AI model group (Experimental): Use the AI-model to locate kidney and tumour, assisting surgeon with the operation
  Interventions: Procedure: an AI-based real-time image-guided kidney model system

INTERVENTIONS:
Procedure: an AI-based real-time image-guided kidney model system — Use the AI-model to locate kidney and tumour, assisting surgeon with the operation
  Arms: AI model group

SUMMARY:
The goal of this study is to develop a real-time artificial intelligence-driven 3D kidney model to assist robotic or laparoscopic partial nephrectomy:

• Can this AI-powered model optimize the workflow of partial nephrectomy and enhance surgical benefits?

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of the AI-based real-time image-guided kidney model system in optimizing partial nephrectomy workflows. Patients scheduled for laparoscopic or robotic-assisted partial nephrectomy will be randomized to receive either AI-assisted surgical navigation (utilizing intraoperative 3D model overlay with automated registration) or conventional approaches. Comparative metrics will include ischemia time, margin positivity rate, and operative efficiency indices. Findings will inform iterative refinement of the system architecture based on clinical performance feedback.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years, regardless of gender
* Written informed consent obtained from the patient or legally authorized representative after full protocol disclosure
* Preoperative imaging (CT/MRI) confirming clinical stage T1a or select T1b renal tumors suitable for partial nephrectomy (R.E.N.A.L. nephrometry score ≤10)
* Localized renal tumors without lymph node/distant metastasis per NCCN Guidelines® (v2023)
* Elective minimally invasive partial nephrectomy (laparoscopic/robotic) after comprehensive surgical counseling

Exclusion Criteria:

* Multifocal renal tumors (bilateral or unilateral)
* Prior systemic anticancer therapy (targeted agents/immunotherapy/chemotherapy) within 6 months
* Absolute surgical contraindications (e.g., ASA class ≥IV, uncontrolled coagulopathy)
* Intraoperative conversion to radical nephrectomy or open approach
* Postoperative adjuvant therapy during protocol-defined follow-up (12 months)
* Major comorbidities (e.g., NYHA class III/IV heart failure, eGFR <30 mL/min/1.73m²) affecting outcome assessment
* Concurrent enrollment in interventional clinical trials
* Investigator-determined ineligibility based on risk-benefit analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Operative Time | Intraoperative

SECONDARY OUTCOMES:
Operating Surgeon's Assessment | immediately after the surgery
  Scoring for Each Surgery(0-5) by navigation accuracy, image rendering smoothness

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), Nanjing, Jiangsu, China